CLINICAL TRIAL: NCT05510284
Title: Post-partum Care in the NICU
Acronym: PeliCaN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Heather Burris, Associate Professor of Pediatrics, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 851606
Record Dates: First submitted 2022-08-17; First posted 2022-08-22 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Postpartum Period

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doula Coordinated-Care Arm (Active Comparator): Postpartum care will be doula-coordinated. The doula will meet with the mother at least once a week during their infant's NICU stay, with a minimum of 3 meetings. Participants will be given the option of seeing the study nurse midwife or their own provider. If the participant opts to see the nurse midwife, they can meet in a private office located in the NICU. The doula, as typical of the doula role, will coordinate any needed community services in the transition to home.
  Interventions: Other: Doula-coordinated, midwife-delivered postpartum care
- Standard Postpartum Care Arm (No Intervention): In this arm participants will receive usual postpartum care. They will be discharged from the hospital while their baby is still in the NICU and a plan will be made to for follow-up with their provider as an outpatient at some point in the next 6 weeks. The study coordinator will provide the participant with a community postpartum resources list.

INTERVENTIONS:
Other: Doula-coordinated, midwife-delivered postpartum care — A doula will coordinate all postpartum care and provide support to the participant. A midwife will be available on-site in the NICU to provide postpartum care.
  Arms: Doula Coordinated-Care Arm

SUMMARY:
This is a pilot randomized control trial to demonstrate the feasibility of a novel model of dyad-centered, doula-coordinated, midwife-delivered postpartum care located in the NICU in a large urban hospital.

ELIGIBILITY:
Inclusion Criteria:

* Preterm birth <34 weeks
* Signed medical record release form

Exclusion Criteria:

* Unable to read or sign informed consent
* If the medical team believes that the infant may die or be transferred to another hospital in upcoming weeks
* PI Discretion

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
Time to receipt of postpartum care | birth until 6 weeks post-partum
  To be analyzed using a wilcoxin rank sum test

SECONDARY OUTCOMES:
Comparison of effectiveness of intervention for mothers with public vs private insurance | birth until 6 weeks post-partum
  Time to receipt of postpartum care will be compared between mothers with public vs private insurance
Comparison of effectiveness of intervention for mothers with infants less than 29 weeks gestational age vs those 29 weeks or older. | birth until 6 weeks post-partum
  Time to receipt of postpartum care will be compared between mothers with infants with a gestational age of less than or equal to 28 6/7 weeks vs a gestational age greater than or equal to 29 weeks
Receipt of Postpartum care | birth until 6 weeks post-partum
  Binary (yes/no), fishers exact test

OTHER OUTCOMES:
Health related quality of life measured by the CDC Health-Related Quality of Life (HRQOL) | 6 months postpartum
  A 14 item survey scoring between 0 and 30, in which a higher score represents a worse health related quality of life
Depression measured by the Edinburgh Postnatal Depression Scale | 6 months postpartum
  Scored 0 through 30, with 30 indicating a worse outcome
Health care utilization - Number of visits | Time of birth until 6 months postpartum
  PhenXToolkit- 270101 Heathcare utilization and access survery
Breastfeeding- ever | 6 months postpartum
  PhenXToolkit-50101 BreasfeedingOutcomes: ever received breastmilk
Breastfeeding- length of time exclusive breastmilk | 6 months postpartum
  PhenXToolkit-50101 BreasfeedingOutcomes: length of time exclusive breastmilk
Breastfeeding- age at stopping breastmilk | 6 months postpartum
  PhenXToolkit-50101 BreasfeedingOutcomes:age at stopping breastmilk receipt (if relevant))
Diet | 6 months postpartum
  Dietary Screener Questionaire (DSQ) 30-items NHANES (Outcome: Cups of fruits or vegetables per day, [more is better])
Physical activity | 6 months postpartum
  International physical activity questionnaire - short form (Scored as Total physical activity, expressed as minutes per week)
Posttraumatic stress disorder symptoms (PTSD) | 6 months postpartum
  PTSD Checklist for DSM-5 (PCL-5), Scored 0 to 40 with a 40 indicating a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No